CLINICAL TRIAL: NCT00394875
Title: The Diabetes Specialist Nurse as Delegated Main Care Provider for Patients With Type 2 Diabetes in a Secondary Care Setting: a Randomized Controlled Trial.
Brief Title: The Diabetes Specialist Nurse as Delegated Main Care Provider for Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Research Foundation, The Netherlands (Other)
Collaborators: Netherlands: Ministry of Health, Welfare and Sports (Other Government); Langerhans Foundation, the Netherlands (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IC-06-03-SL
Record Dates: First submitted 2006-10-31; First posted 2006-11-02 (Estimated); Last update posted 2006-11-02 (Estimated); Status verified 2006-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Randomized controlled trial; Delegation, Professional; Nurses
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Therapeutics

INTERVENTIONS:
Procedure: Treated and educated by nurses specialized in diabetes.

SUMMARY:
To determine whether the management of type 2 diabetes mellitus (DM2) can be transferred from an internist to a supervised nurse specialized in diabetes (NSD) with a comparable quality of clinical care, health care costs, health related quality of life (HRQOL), and patient satisfaction.

DETAILED DESCRIPTION:
Diabetes mellitus type 2 (DM2) is a chronic, progressive illness which causes considerable morbidity and premature mortality.1-2 The worldwide prevalence of DM2 is high and is increasing steadily, also in The Netherlands.3-4 The burden of DM2 on health care has also increased because of the intensified cardiovascular risk management being practiced to prevent macrovascular morbidity and mortality in these patients.5 In the treatment of DM2, tight guidelines are increasingly recommended for optimizing glycaemia, blood pressure and lipid profile.6 Therefore, the burden of treatment has increased and will further increase per patient as well as per population with DM2. In order to meet this problem, we tested, in the current study, the hypothesis that well defined routine aspects in diabetes care, previously handled only by medical doctors in secondary care setting, may be safely transferred to supervised nurses specialized in diabetes (NSD), including the prescription of medication, resulting in at least the same quality of clinical care, health care costs, health related quality of life (HRQOL), and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* patients with DM2 who were referred by GPs to the diabetes outpatient clinics

Exclusion Criteria:

* macroalbuminuria
* serum creatinine level > 135 mol/l,
* Cockcroft < 50 ml/min
* alanine aminotransferase (ALT) > 120 U/l
* pregnant woman

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81
Dates: Start 2002-03; Study Completion 2005-01

PRIMARY OUTCOMES:
mean decrease in:
HbA1c
blood pressure
total cholesterol
LDL cholesterol
cholesterol/HDL-ratio
proportion of patients achieving ranges of:
glycaemic control
lipid profile

SECONDARY OUTCOMES:
health related quality of life (HRQOL)
diabetes related symptoms
patients' satisfaction
health care consumption and costs

CONTACTS AND LOCATIONS:
Overall Officials: Sebastiaan T Houweling, PhD, Principal Investigator — 2. Department of General Practice, University of Groningen, Groningen, The Netherlands; Betty Meyboom-de Jong, PhD, Study Chair — Department of General Practice, University of Groningen, Groningen, The Netherlands; Henk Bilo, PhD, Study Chair — 3. Centre of Excellence, Isala Clinics, Zwolle, The Netherlands
Locations (1):
- Isala Clinics, Zwolle, Netherlands